CLINICAL TRIAL: NCT03877848
Title: EluNIR Ridaforolimus Eluting Coronary Stent System in Patients at High Bleeding Risk (HBR)- EluNIR HBR Study
Status: Completed | Type: Observational
Sponsor: Medinol Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: EluNIR HBR study
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Coronary Stenosis
Keywords: bleeding; PCI
MeSH Terms: conditions — Coronary Stenosis; Hemorrhage | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- ACS and Non-ACS: DAPT will be stopped at 30 days in non-ACS subjects while at ACS Patients it may be maintained for up to 3 months. In patients with ACS or with an ischemic event during the first 30 days, DAPT may be continued at the discretion of the investigator. In ACS patients DAPT should be continued for a maximum of 3 months. For patients with recurrent ischemic events duration of DAPT therapy will be at the discretion of the investigator.
  Patients receiving long-term oral anticoagulation with either a Vitamin K inhibitor or a NOAC/DOAC will receive either single antiplatelet therapy with clopidogrel, or DAPT for 30 days (triple therapy) followed by single antiplatelet therapy with clopidogrel. Clopidogrel (75 mg QD) will be given to these patients post procedure for 6 months in stable patients and 12 months in ACS patients.
  Interventions: Device: Percutaneous Coronary Intervention (PCI)

INTERVENTIONS:
Device: Percutaneous Coronary Intervention (PCI) — Patients enrolled to the study will undergo angiography followed by PCI according to current guidelines.

SUMMARY:
The study will enroll approximately 316 subjects with a wide spectrum of PCI indications (stable angina as well as ACS), who are considered to be at high risk of bleeding. Patients will undergo PCI with implantation of the EluNIR stent, followed by shortened duration (1 months in stable patients, and up to 3 months in ACS patients) of DAPT.

DETAILED DESCRIPTION:
This is a prospective, multi-center (Up to 20 sites), single-arm, open-label post marketing clinical trial.

The objectives: To assess the safety and efficacy of shortened DAPT duration (30 days in stable patients and up to 90 days in ACS patients) following PCI using the EluNIR stent, in patients considered to be at high bleeding risk (HBR).

Patients will be enrolled to the study prior to the PCI procedure.Once a patient has signed an informed consent, met all general and angiographic eligibility criteria, and a guidewire has successfully been passed beyond the target lesion and lesion preparation (if indicated) completed, the patient will be enrolled into the trial.Data collection commences after the subject has signed the informed consent form. Data collection including subject demographic information, laboratory tests, and procedural data as well as follow-up visits or telephone contacts will be captured by the Investigator or site coordinator who has been trained on the CIP and Case Report Forms (CRF).

After discharge from the hospital, each subject will be followed with an in-clinic follow-up visit at 30 days, and follow-up by phone at 6 months and 1year post procedure. Patients with recurrent ischemic events within the first 30 days as well as patients in whom the initial presentation was ACS and in whom the investigator has decided to continue DAPT beyond 30 days will have an additional phone follow-up at 3 months.

The clinical investigation will last for the expected duration of each subject's participation.

Each subject will remain in the clinical investigation for approximately 1 year from the time of the study stent implantation until the last follow-up telephone contact.

The trial population will consist of approximately 316 male and female subjects undergoing PCI for angina (stable or unstable), silent ischemia, non-ST elevation MI (NSTEMI) considered at HBR.

ELIGIBILITY:
Inclusion Criteria:

All inclusion criteria must be present for the patient to be eligible for enrollment.

General Inclusion Criteria

1. Age ≥ 18 years.
2. Patient with angina (stable or unstable), silent ischemia or NSTEMI, undergoing PCI using the EluNIR stent.
3. Patient or legal guardian is willing and able to provide informed written consent and comply with follow-up visits and testing schedule.

In addition, patients must meet at least one of the following criteria for high risk of bleeding:

1. Age ≥75 years
2. Oral anticoagulation planned to continue after PCI
3. Hemoglobin <11 g/liter or anemia requiring transfusion within 12 weeks before enrollment to the study
4. Platelet count< 100,000/mm³
5. Hospital admission for bleeding in previous 12 months
6. Stroke in previous 12 months
7. Previous intracerebral hemorrhage
8. Severe chronic liver disease defined as patients who have developed any of the following: variceal hemorrhage, ascites, hepatic encephalopathy or jaundice
9. Renal failure defined as creatinine clearance< 40 ml/min
10. Non-skin cancer diagnosed or treated < 3 years
11. Planned surgery within 12 months that would require interruption of DAPT
12. Planned daily NSAID (other than aspirin) or steroids for > 30 days after PCI
13. Expected nonadherence to >30 days of dual antiplatelet therapy in stable patients and >3 months in ACS patients

Angiographic inclusion criteria (visual estimate)

1. Complex lesions are allowed including calcified lesions (lesion preparation with scoring/cutting and rotational atherectomy are allowed), presence of thrombus that is non-occlusive and does not require thrombectomy, CTO, bifurcation lesions (except planned dual stent implantation), ostial RCA lesions, tortuous lesions, bare metal stent restenotic lesions, protected left main lesions, and saphenous vein graft lesions.
2. Up to 2 overlapping stents are allowed (ie, one overlap)

Exclusion Criteria:

All exclusion criteria must be absent for the patient to be eligible for enrollment.

General Exclusion Criteria

1. Pregnant and breastfeeding women
2. Patients requiring a planned staged PCI with a non-study stent
3. Patients expected not to comply with 1-month DAPT.
4. Patients expected not to comply with long-term single anti-platelet therapy
5. PCI during the previous 12 months with a non-study stent
6. History of stent thrombosis
7. Cardiogenic shock (defined as persistent hypotension (systolic blood pressure <90 mm/Hg for more than 30 minutes) or requiring pressors or hemodynamic support, including IABP.
8. Subject is intubated.
9. Known LVEF <30%.
10. White blood cell (WBC) count <3,000 cells/mm3.
11. Active bleeding from any site at time of inclusion
12. Known allergy to protocol-required concomitant medications such as aspirin, or DAPT (clopidogrel, prasugrel, ticagrelor), or heparin and bivalirudin, or iodinated contrast that cannot be adequately pre-medicated.
13. Any co-morbid condition that may cause non-compliance with the protocol (e.g. dementia, substance abuse, etc.) or reduced life expectancy to <12 months (e.g. cancer, severe heart failure, severe lung disease).
14. Patient has received an organ transplant or is on a waiting list for an organ transplant.
15. Participation in another clinical trial that has not reached its primary endpoint.

Angiographic Exclusion Criteria (visual estimate)

1. Visually estimated RVD<2.5 mm or >4.25mm.
2. Unprotected left main intervention.
3. Ostial LAD and/or LCx intervention
4. Bifurcation lesions with dual stent implantation.
5. Stenting of lesions due to DES restenosis.
6. Total stented length > 60 mm
7. Planned implantation of any DES which is not EluNIR

Note: In case the procedure required the unplanned implantation of a different (non-EluNIR) stent the subject will be de-registered from the study.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High bleeding risk subjects undergoing PCI using the EluNIR stent for angina, silent ischemia or non STEMI.
Sampling Method: Non-Probability Sample
Enrollment: 319 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
The composite of cardiac death, myocardial infarction, or stent thrombosis at 1 year (ARC definite and probable) | 1 Year

SECONDARY OUTCOMES:
TLF, defined as the composite of cardiac death, target vessel-related MI, or ischemia-driven TLR. | To be evaluated at 30 days, 6 months, and 1 year
Major adverse cardiac events (MACE; the composite rate of cardiac death, any MI or ischemia-driven TLR) | To be evaluated at 30 days, 6 months, and 1 year
Target vessel failure (TVF; the composite rate of death, target vessel related MI or ischemia-driven TVR) | To be evaluated at 30 days, 6 months, and 1 year
The composite of cardiac death, myocardial infarction, or stent thrombosis at 30 days and 6 months | To be evaluated at 30 days, 6 months, and 1 year
All-cause mortality | To be evaluated at 30 days, 6 months, and 1 year
Cardiac death | To be evaluated at 30 days, 6 months, and 1 year
Bleeding events according to BARC definitions | To be evaluated at 30 days, 6 months, and 1 year
Myocardial Infarction | To be evaluated at 30 days, 6 months, and 1 year
Target Vessel Related MI | To be evaluated at 30 days, 6 months, and 1 year
Ischemia-driven TLR | To be evaluated at 30 days, 6 months, and 1 year
Ischemia-driven TVR | To be evaluated at 30 days, 6 months, and 1 year
Stent Thrombosis (ARC definite and probable) | To be evaluated at 30 days, 6 months, and 1 year
Bleeding complications (BARC definitions), evaluated as components and as a composite of BARC Type 3 and 5 bleeding | To be evaluated at 30 days, 6 months, and 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Medinol LTD, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kornowski R, Konigstein M, Jonas M, Assali A, Vaknin-Assa H, Segev A, Danenberg H, Halabi M, Roguin A, Kerner A, Lev E, Karamasis GV, Johnson TW, Anderson R, Blaxill J, Jadhav S, Hoole S, Witberg G, Issever MO, Ben-Yehuda O, Baumbach A. Percutaneous Coronary Interventions Using a Ridaforolimus-Eluting Stent in Patients at High Bleeding Risk. J Am Heart Assoc. 2024 Jan 16;13(2):e029051. doi: 10.1161/JAHA.122.029051. Epub 2024 Jan 12. PMID 38214256